CLINICAL TRIAL: NCT00439699
Title: A Pilot Clinical Trial of Memantine for Essential Tremor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: Ralph M. Parsons Foundation (Other); Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Adrian Handforth, MD, Assistant Chief, Neurology, VAMC, VA Greater Los Angeles Healthcare System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0033
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Memantine; Clinical Trial
MeSH Terms: conditions — Essential Tremor | interventions — Memantine

ARMS (1):
- Memantine (Experimental): Tremor reduction
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Mematine administration

SUMMARY:
The purpose of this study is to obtain information on whether or not the medication Memantine reduces tremor in persons with essential tremor and is well-tolerated.

DETAILED DESCRIPTION:
Background: Essential tremor (ET) is the most common movement disorder but has relatively few effective and tolerated therapies. Tremor in ET is believed to be generated by a central oscillator, the inferior olivary nucleus. Membrane potentials in neurons of this nucleus oscillate at tremor frequency. Evidence indicates that the ability of this nucleus to produce tremor is medicated by glutamate acting on the NMDA receptor. As NMDA receptor antagonists suppress tremor, it is suggested that memantine, a low affinity NMDA antagonist, will be effective for essential tremor.

Objective: To assess the efficacy, safety and stability of response to memantine in a pilot single-site feasibility rising-dose trial in the treatment of essential tremor.

Method: Subjects with bilateral upper extremity essential tremor, on no essential tremor therapy, or on a stable-dose therapy, will have laboratory tests and EKG tests at a screening visit. Eligible subjects will have baseline tremor assessments with standardized rating scales. The tremor will be videotaped. In the first titration step, all subjects will take memantine at the dose of 5 mg/day for 2 weeks, then 5 mg twice a day for another 2 weeks, and tremor again assessed. In the second titration step the dose will similarly be raised to 20 mg/day, taken as 10 mg twice a day, and tremor assessed 4 weeks after the last tremor assessment. In the third titration step, the dose will be raised to 30 mg/day, taken as 15 mg twice a day, and tremor assessed at the conclusion of the third titration step. In the fourth titration step, the dose will be raised to 40 mg/day, taken as 20 mg twice a day, and tremor assessed at the conclusion of the fourth titration step. The dose will be adjusted downwards if titration is not tolerated. Subjects who achieve a clinically meaningful tremor reduction will enter a 12-week extension study assessing the stability of the tremor response.

Data analysis: Subjects will be recruited according to a two-part Gehan design. A "responder" is defined as a 30% reduction in the tremor score. To assess whether memantine has a potential responder rate of 30 percent, 9 subjects will be recruited in the first phase. If at least one subject is a responder, another 16 subjects will be recruited to estimate the actual responder rate with a standard error of 10%.

Conclusions: If memantine is effective in suppressing tremor, it would be welcomed by patients and the movement disorders community as a well-tolerated new treatment for essential tremor.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Subject diagnosed with essential tremor affecting both upper extremities.
* Subject has been diagnosed for at least one year with tremor that is troublesome, so that improvement of tremor would improve the quality of life.
* Subject has tremor with a tremor rating scale severity of 2 to 4 in one or both upper extremities in the tremor rating scale during posture and/or kinesis.
* Subject has not had satisfactory tremor response to at least one anti-tremor medication.
* Subject is able to comply with all testing and follow-up visit requirements.
* Subject is able to abstain from alcohol for at least 12 hours prior to each Study Visit and from caffeinated beverages on the day of the Visit.
* Subject has voluntarily signed an informed consent in accordance with institutional policies.
* Subject is either

  * Not taking medication for Essential Tremor and has not done so for at least 28 days prior to Visit 1.
  * Taking medication for Essential Tremor and has been taking a stable dose so for at least 28 days prior to Visit 1.

Exclusion Criteria:

* Subject has progressive neurological disease other than Essential Tremor.
* Subject has history of alcoholism or drug abuse within the past year.
* Subject has history of mania, bipolar depressive disorder, schizophrenia, or other major psychiatric disorder.
* Subject drinks more than 2 glasses of wine or equivalent per day in last 30 days.
* Subject has received botulinum injection of the upper extremities in the past 6 months.
* Subject is currently using investigational device.
* Subject has taken an investigational drug within a clearance duration of 5 times the half-life of the investigational drug.
* Subject is pregnant or a female of childbearing potential not using adequate contraception.
* Subject has a medical condition likely to result in hospitalization.
* Known allergy to memantine or amantadine.
* Taking medication that alkalinizes the urine, such as carbonic anhydrase inhibitor or sodium bicarbonate.
* Any disorder or condition that may interfere with the absorption, the distribution, or excretion of drugs.
* Taking medication known to cause postural tremor, that in the clinical judgement of the investigator is contributing to the subject's tremor.
* Receiving deep brain stimulation within two weeks prior to Visit 1 or has potential need for deep brain stimulation during the study.
* Has received ablative thalamotomy or gamma knife thalamotomy within six months of study onset.
* Tremor potentially due to head trauma, hyperthyroidism, cerebrovascular disease, multiple sclerosis, polyneuropathy, or family history of Fragile X syndrome.
* Known renal disease with creatinine level outside normal range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The degree of tremor at the end of the dose adjustment phase compared to baseline | Six months

SECONDARY OUTCOMES:
Quality of Life. | Six months
Degree of tremor at the end of the extension phase compared to the beginning of the extension phase. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Handforth, M.D., Principal Investigator — Veteran Affairs Greater Los Angeles
Locations (1):
- VA Greater Los Angeles, Los Angeles, California, United States